CLINICAL TRIAL: NCT00725309
Title: Specialized Center of Clinically Oriented Research: Alveolar and Airway Mechanisms for COPD: Genetic Determinants: Elastin Quality and Quantity (Project 2)
Brief Title: Evaluating Genetic Factors That May Contribute to Elastin Function and the Development of Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 576 -201108294
Record Dates: First submitted 2008-07-29; First posted 2008-07-30 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Emphysema; Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Obstructive Pulmonary Disease; COPD; Elastin; ELN
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive; Aortic Stenosis, Supravalvular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma, serum, isolated RNA and DNA, lung tissue (obtained from other substudies)
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a lung disease that is primarily caused by cigarette smoking. The breakdown of elastin, a protein found in the lungs, can cause lung damage and may contribute to the development of COPD. Some people may be more prone to elastin damage and in turn to developing COPD than others. This study will examine whether genetic factors are responsible for altering elastin function and increasing the risk of developing COPD.

DETAILED DESCRIPTION:
COPD is a disease in which the lung airways are damaged and partly obstructed, making it difficult to breathe. There is no cure for this disease, and it is the fourth leading cause of death in the United States. Symptoms include coughing, excess mucus production, shortness of breath, wheezing, and chest tightness. The most common risk factor for developing COPD is cigarette smoking; however, only 15% to 20% of smokers are diagnosed with COPD in their lifetimes, suggesting that some smokers are more prone to developing COPD than others. Elastin, a protein found in the tissues surrounding the lung airways and in the alveolar walls of the lung, is essential for healthy lung function. As elastin breaks down, lung damage can occur, potentially leading to COPD. It is thought that some people may be genetically predisposed to elastin damage by cigarette smoke, thus accounting for the select group of smokers affected by COPD. This study will examine the ways in which elastin defects contribute to the development of COPD. Researchers will examine whether genetic variations play a role in altering elastin function and in influencing health outcomes in people with COPD.

This study will enroll people with COPD that was caused by emphysema. Participants will complete one study visit that will include a medical record and history review and blood collection (or saliva collection, if blood draw is unsuccessful). A portion of blood will be stored for future genetic research. Participants will also complete questionnaires to collect information on activities, health, and quality of life. Study researchers will contact participants at the end of the study to collect follow-up medical information.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 18 years
* Ability to read and write in English
* Able to participate in the informed consent process
* Acceptable pulmonary function tests (PFTs) done at Barnes-Jewish Hospital within 1 month of study enrollment
* Relatively stable clinical status (not experiencing COPD exacerbation in the previous 6 weeks)
* Global Initiative for Chronic Obstructive Lung Disease (GOLD) class III or IV COPD (FEV1/FVC less than 70% and FEV1 less than 50% of predicted value)

Exclusion Criteria:

* Pregnant
* Prisoner
* Vulnerable populations
* Pi Z phenotype (i.e., alpha-1 antitrypsin deficiency)
* Significant lung disease, other than COPD / emphysema / chronic bronchitis (e.g., interstitial lung disease, asthma or other predominant airway disease, cystic fibrosis, active tuberculosis)
* Known active hepatitis B, hepatitis C, or HIV/AIDS (found in medical record review; not prospectively evaluated)
* Coexisting active chronic inflammatory or collagen vascular disease, immunodeficiency of any kind, non-cutaneous malignancy (melanoma is an exclusion), or previous organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll people who undergo evaluation or follow-up at Barnes-Jewish Hospital for lung volume reduction surgery (LVRS). Researchers will also enroll eligible COPD patients from other Washington University Medical Center pulmonary clinics.
Sampling Method: Non-Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2007-11; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert P. Mecham, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States